CLINICAL TRIAL: NCT06690996
Title: A Phase 1, Randomized, Placebo-controlled, Investigator and Participant Blinded, Single-ascending Dose and Multiple-ascending Dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of LY4005130 in Healthy Participants.
Brief Title: A Study of LY4005130 in Healthy Participants
Acronym: FPAB
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 27231; J5D-MC-FPAB (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- LY4005130 Part A (SAD) SC (Experimental): A single-ascending dose of LY4005130 administered subcutaneously (SC)
  Interventions: Drug: LY4005130
- Placebo Part A (SAD) SC (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo
- LY4005130 Part A (SAD) IV (Experimental): A single-ascending dose of LY4005130 administered intravenously (IV)
  Interventions: Drug: LY4005130
- Placebo Part A (SAD) IV (Placebo Comparator): Placebo administered IV
  Interventions: Drug: Placebo
- LY4005130 Part A (SAD) Optional (Experimental): A single-ascending dose of LY4005130 administered either SC or IV depending on emerging data from earlier cohorts
  Interventions: Drug: LY4005130
- Placebo Part A (SAD) Optional (Placebo Comparator): A single-ascending dose of placebo administered either SC or IV depending on emerging data from earlier cohorts
  Interventions: Drug: Placebo
- LY4005130 Part B (MAD) IV (Experimental): Multiple-ascending doses of LY4005130 administered IV
  Interventions: Drug: LY4005130
- Placebo Part B (MAD) IV (Placebo Comparator): Placebo administered IV
  Interventions: Drug: Placebo
- LY4005130 Part B (MAD) SC or IV (Experimental): Multiple-ascending doses of LY4005130 administered either SC or IV depending on emerging data from earlier cohorts
  Interventions: Drug: LY4005130
- Placebo Part B (MAD) SC or IV (Placebo Comparator): Multiple-ascending doses of placebo administered either SC or IV depending on emerging data from earlier cohorts
  Interventions: Drug: Placebo
- LY4005130 Part B (MAD) Optional (Experimental): Multiple-ascending doses of LY4005130 administered either SC or IV depending on emerging data from earlier cohorts
  Interventions: Drug: LY4005130
- Placebo Part B (MAD) Optional (Placebo Comparator): Multiple-ascending doses of placebo administered either SC or IV depending on emerging data from earlier cohorts
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY4005130 — Administered IV
  Arms: LY4005130 Part A (SAD) IV; LY4005130 Part A (SAD) Optional; LY4005130 Part B (MAD) IV; LY4005130 Part B (MAD) Optional; LY4005130 Part B (MAD) SC or IV
Drug: LY4005130 — Administered SC
  Arms: LY4005130 Part A (SAD) Optional; LY4005130 Part A (SAD) SC; LY4005130 Part B (MAD) Optional; LY4005130 Part B (MAD) SC or IV
Drug: Placebo — Administered IV
  Arms: Placebo Part A (SAD) IV; Placebo Part A (SAD) Optional; Placebo Part B (MAD) IV; Placebo Part B (MAD) Optional; Placebo Part B (MAD) SC or IV
Drug: Placebo — Administered SC
  Arms: Placebo Part A (SAD) Optional; Placebo Part A (SAD) SC; Placebo Part B (MAD) Optional; Placebo Part B (MAD) SC or IV

SUMMARY:
The purpose of this study is to evaluate how well LY4005130 is tolerated and what side effects may occur in healthy participants. The study drug will be administered either subcutaneously (SC) (under the skin) or intravenously (IV) (into a vein in the arm). Blood tests will be performed to check how much LY4005130 gets into the bloodstream and how long it takes the body to eliminate it.

Part A for the single-ascending doses (SAD) of the study will last about 12 weeks with 9 visits. Part B for the multiple-ascending doses (MAD) of the study will either last about 16 weeks with 13 visits or 26 weeks with 14 visits not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs, and 12-lead (electrocardiogram) ECG. If any values are outside the normal range and considered to be significant, for example, elevated white blood cell count, the respective test may be repeated once at the discretion of the investigator without consultation with the sponsor
* If enrolled as Japanese or Chinese, the entry requirements are as follows:

  * To qualify as a participant of first-generation Japanese origin, the participant, the participant's biological parents, and all of the participant's biological grandparents must be of exclusive Japanese descent and born in Japan
  * To qualify as Chinese for the purpose of this study, all 4 of the participant's biological grandparents must be of exclusive Chinese descent and born in China
* Have a body weight 45 kilogram (kg) or greater and body mass index greater than 18 and less than 32 kilogram per square meter (kg/m²)

Exclusion Criteria:

* Are an individual of childbearing potential (IOCBP)
* Have known allergies to LY4005130, related compounds, or any components of the formulation
* Have received a live vaccine within 28 days of screening or intend to do so during the study or within 28 days after the study

  * Non-live or inactivated vaccinations are allowed
  * Bacillus Calmette Guerin vaccine must not have been administered within 12 months before screening
* Had a surgical procedure within 12 weeks before screening;

  * during the study, or
  * within 28 days after the study
* Have a history of allergy to medications that could be used to treat infusion reactions, or to the drug excipients
* Have a history or presence of multiple or severe allergies, anaphylactic reaction to prescription or nonprescription drugs, significant history of atopy, or a history of severe posttreatment hypersensitivity reactions. These reactions include, but are not limited to, erythema multiforme major, linear immunoglobulin A dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis
* Have a diagnosis or history of malignant disease within 5 years prior to screening, with the following exceptions

  * Basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years, or
  * Cervical carcinoma in situ, with no evidence of recurrence within the 5 years prior to screening
* Have had breast cancer within the past 10 years
* Have a history of a primary immunodeficiency, splenectomy, or any underlying condition that predisposes the participant to infection that, in the opinion of the sponsor or investigator, poses an unacceptable risk to the participant
* Have a current or recent acute, active infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline to Study Completion (Up to 26 Weeks)
  A summary of TEAEs and SAEs regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY4005130 | Baseline to Study Completion (Up to 26 Weeks)
  Cmax of LY4005130
PK: Area Under the Concentration Versus Time Curve (AUC) of LY4005130 | Baseline to Study Completion (Up to 26 Weeks)
  AUC of LY4005130

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Fortrea Clinical Research Unit, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No